CLINICAL TRIAL: NCT07101367
Title: A Comparative Study Between Dexmedetomidine Versus Methylprednisolone on Induced Inflammatory Response in Patients Undergoing On-pump CABG
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: FMASU MD219/2023
Record Dates: First submitted 2025-07-24; First posted 2025-08-03 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2024-08

CONDITIONS: Coronary Artery Disease; Systemic Inflammatory Response Syndrome; Postoperative Complications
MeSH Terms: conditions — Coronary Artery Disease; Systemic Inflammatory Response Syndrome; Postoperative Complications | interventions — Saline Solution; Control Groups; Dexmedetomidine; Methylprednisolone; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Intervention Model Description: Control group without any medications Dexmedetomidine group Methylprednisolone group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized Double blinded clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Control (Active Comparator): Control group receiving 10 ml of normal saline after induction of anesthesia then followed by infusion of normal saline till extubation in ICU
  Interventions: Drug: Normal saline
- Dexmedetomidine (Active Comparator): Starting with precedex loading dose after anesthesia induction then infusion till extubation in ICU
  Interventions: Drug: Dexmedetomidine
- Methylprednisolone (Active Comparator): To be diluted in 10 ml normal saline then given after induction of anesthesia then followed by normal saline infusion till extubation in ICU
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Normal saline — After induction of anesthesia give 10 ml of normal saline then followed by infusion of normal saline till extubation of patient in ICU
  Other Names: Control group (placebo)
  Arms: Control
Drug: Dexmedetomidine — After induction of anesthesia give loading dose of precedex 1 mcg/kg diluted in 10 ml normal saline then attach syringe pump of precedex infusion of 0.5mcg/kg/hr till extubation in ICU
  Other Names: Precedex (active comparator)
  Arms: Dexmedetomidine
Drug: Methylprednisolone — After induction of anesthesia give solumedrol of a dose 10mg/kg diluted in 10ml of normal saline followed by a normal saline infusion till the extubation of the patient in the ICU
  Other Names: Solumedrol (active comparator)
  Arms: Methylprednisolone

SUMMARY:
A comparison between precedex versus solumedrol as anti-inflammatory stress response inhibitors in patients undergoing on-pump CABG using different inflammatroy response parameters and the outcome of the drugs on the cognitive and cardiac status post extubation

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-60 years.
2. Sex: Both sexes.
3. American Society of Anaesthesiologists (ASA) Physical Status Class II, and III.
4. Scheduled for CABG on cardio-pulmonary bypass.

Exclusion Criteria:

1. Declining to give a written informed consent.
2. History of allergy to the medications used in the study.
3. Psychiatric disorders.
4. Significant cognitive dysfunction.
5. American Society of Anesthesiologists (ASA) Physical Status Class IV.
6. Chronic liver or kidney disease.
7. Poor systolic function ( Ejection fraction < 40% ).
8. Pregnancy.
9. Redo CABG.

9.Infection during the week preceding surgery white blood cell count over 11,000 mm3 10.Pre-operative use of antibiotics or corticosteroids.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Induced inflammatory response | First 24 hours post cardio-pulmonary bypass
  Effect of both drugs on attenuating induced inflammatory response

SECONDARY OUTCOMES:
Cognitive function | First 24 hours post cardio-pulmonary bypass
  Assesment of post operative cognitive function and occurnce of post operative delerium using CAM-ICU score

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Cairo Governorate, Egypt